CLINICAL TRIAL: NCT02460887
Title: A Randomized Trial Comparing Induction Gemcitabine and Cisplatin Plus Intensity-modulated Radiotherapy with Concurrent Cisplatin Plus Intensity-modulated Radiotherapy in Patients with Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: The Role of Induction Gemcitabine and Cisplatin in Locoregionally Advanced Nasopharyngeal Carcinoma in the Era of IMRT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Yu Huang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sun Yat-sen University HPY
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Induction chemotherapy+IMRT gemcitabine and cisplatin regimen Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 2 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT).
  Interventions: Drug: Gemcitabine; Drug: cisplatin; Radiation: Intensity-modulated Radiotherapy
- Active Comparator (Active Comparator): IMRT and concurrent cisplatin Patients receive intensity modulated-radiotherapy (IMRT), concurrently with weekly cisplatin 40 mg/m² up to 7cycles.
  Interventions: Drug: cisplatin; Radiation: Intensity-modulated Radiotherapy

INTERVENTIONS:
Drug: Gemcitabine — Experimental arm: Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 2 cycles before IMRT.
  Arms: Experimental
Drug: cisplatin — Experimental arm: Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 2 cycles before IMRT.
  Other Names: DDP
  Arms: Experimental
Drug: cisplatin — Active Comparator arm: Patients receive weekly cisplatin 40 mg/m² up to 7cycles during IMRT.
  Other Names: DDP
  Arms: Active Comparator
Radiation: Intensity-modulated Radiotherapy — Intensity modulated-radiotherapy (IMRT) is given as 2.0-2.33 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor.
  Other Names: IMRT

SUMMARY:
The purpose of this study is to verify that induction gemcitabine and cisplatin plus intensity-modulated radiotherapy (IMRT) is non-inferior to concurrent weekly cisplatin plus IMRT for patients with locoregionally advanced nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
Patients with non-keratinizing NPC T1-4N2-3或T3-4N0-1M0 (UICC/AJCC 7th edition) are randomly assigned to receive induction chemotherapy or CCRT alone. Patients in experimental group receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 2 cycles before intensity-modulated radiotherapy (IMRT). Patients in control group receive IMRT concurrently with weekly cisplatin 40 mg/m² up to 7cycles.

IMRT is given as 2.0-2.33 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor.

Our primary endpoint is failure-free survival (FFS). Secondary end points include overall survival (OS), locoregional failure-free survival (LR-FFS), distant failure-free survival (D-FFS) rates and toxic effects. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma (including WHO II or III).
* Tumor staged as T1-4N2-3或T3-4N0-1M0 (according to the 7th AJCC edition).
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4000/μL, hemoglobin ≥ 90g/L and platelet count ≥ 100000/μL.
* Adequate liver function: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤1.5×ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 2 years
  Failure-free survival rate is calculated from the date of randomization to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival is calculated from randomization to death from any cause.
Locoregional failure-free survival | 2 years
  Locoregional failure-free survival is calculated from randomization to the first locoregional failure.
Distant failure-free survival | 2 years
  Distant failure-free survival is calculated from randomization to the first remote failure.
Overall response rate | 3 months after completion of IMRT
  Overall response rate at 3 months after completion of IMRT
Number of participants with adverse events | 2 years
  Incidence of acute and late toxicity
Quality of life during treatment | During whole chemotherapy and IMRT treatment.For experimental arm, an expected average of 12 weeks; for active comparator arm, an expected average of 6 weeks.
  Quality of life is measured by FACIT questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yu Huang, M. D., Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Haddad R, O'Neill A, Rabinowits G, Tishler R, Khuri F, Adkins D, Clark J, Sarlis N, Lorch J, Beitler JJ, Limaye S, Riley S, Posner M. Induction chemotherapy followed by concurrent chemoradiotherapy (sequential chemoradiotherapy) versus concurrent chemoradiotherapy alone in locally advanced head and neck cancer (PARADIGM): a randomised phase 3 trial. Lancet Oncol. 2013 Mar;14(3):257-64. doi: 10.1016/S1470-2045(13)70011-1. Epub 2013 Feb 13. PMID 23414589
- [Background] Cohen EE, Karrison TG, Kocherginsky M, Mueller J, Egan R, Huang CH, Brockstein BE, Agulnik MB, Mittal BB, Yunus F, Samant S, Raez LE, Mehra R, Kumar P, Ondrey F, Marchand P, Braegas B, Seiwert TY, Villaflor VM, Haraf DJ, Vokes EE. Phase III randomized trial of induction chemotherapy in patients with N2 or N3 locally advanced head and neck cancer. J Clin Oncol. 2014 Sep 1;32(25):2735-43. doi: 10.1200/JCO.2013.54.6309. Epub 2014 Jul 21. PMID 25049329
- [Background] Fountzilas G, Ciuleanu E, Bobos M, Kalogera-Fountzila A, Eleftheraki AG, Karayannopoulou G, Zaramboukas T, Nikolaou A, Markou K, Resiga L, Dionysopoulos D, Samantas E, Athanassiou H, Misailidou D, Skarlos D, Ciuleanu T. Induction chemotherapy followed by concomitant radiotherapy and weekly cisplatin versus the same concomitant chemoradiotherapy in patients with nasopharyngeal carcinoma: a randomized phase II study conducted by the Hellenic Cooperative Oncology Group (HeCOG) with biomarker evaluation. Ann Oncol. 2012 Feb;23(2):427-35. doi: 10.1093/annonc/mdr116. Epub 2011 Apr 27. PMID 21525406
- [Background] Yi J, Huang X, Gao L, Luo J, Zhang S, Wang K, Qu Y, Xiao J, Xu G. Intensity-modulated radiotherapy with simultaneous integrated boost for locoregionally advanced nasopharyngeal carcinoma. Radiat Oncol. 2014 Feb 18;9:56. doi: 10.1186/1748-717X-9-56. PMID 24533569
- [Background] Zhang L, Zhang Y, Huang PY, Xu F, Peng PJ, Guan ZZ. Phase II clinical study of gemcitabine in the treatment of patients with advanced nasopharyngeal carcinoma after the failure of platinum-based chemotherapy. Cancer Chemother Pharmacol. 2008 Jan;61(1):33-8. doi: 10.1007/s00280-007-0441-8. Epub 2007 Mar 20. PMID 17909810
- [Background] He X, Ou D, Ying H, Zhu G, Hu C, Liu T. Experience with combination of cisplatin plus gemcitabine chemotherapy and intensity-modulated radiotherapy for locoregionally advanced nasopharyngeal carcinoma. Eur Arch Otorhinolaryngol. 2012 Mar;269(3):1027-33. doi: 10.1007/s00405-011-1669-9. Epub 2011 Jun 26. Erratum In: Eur Arch Otorhinolaryngol. 2012 Mar;269(3):1035. Xiayun, He [corrected to He, Xiayun]. PMID 21706324
- [Background] Lee AW, Lau WH, Tung SY, Chua DT, Chappell R, Xu L, Siu L, Sze WM, Leung TW, Sham JS, Ngan RK, Law SC, Yau TK, Au JS, O'Sullivan B, Pang ES, O SK, Au GK, Lau JT; Hong Kong Nasopharyngeal Cancer Study Group. Preliminary results of a randomized study on therapeutic gain by concurrent chemotherapy for regionally-advanced nasopharyngeal carcinoma: NPC-9901 Trial by the Hong Kong Nasopharyngeal Cancer Study Group. J Clin Oncol. 2005 Oct 1;23(28):6966-75. doi: 10.1200/JCO.2004.00.7542. PMID 16192584
- [Background] Chan AT, Teo PM, Ngan RK, Leung TW, Lau WH, Zee B, Leung SF, Cheung FY, Yeo W, Yiu HH, Yu KH, Chiu KW, Chan DT, Mok T, Yuen KT, Mo F, Lai M, Kwan WH, Choi P, Johnson PJ. Concurrent chemotherapy-radiotherapy compared with radiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: progression-free survival analysis of a phase III randomized trial. J Clin Oncol. 2002 Apr 15;20(8):2038-44. doi: 10.1200/JCO.2002.08.149. PMID 11956263
- [Background] Lee AW, Lau KY, Hung WM, Ng WT, Lee MC, Choi CW, Chan CC, Tung R, Cheng PT, Yau TK. Potential improvement of tumor control probability by induction chemotherapy for advanced nasopharyngeal carcinoma. Radiother Oncol. 2008 May;87(2):204-10. doi: 10.1016/j.radonc.2008.02.003. Epub 2008 Mar 10. PMID 18329742
- [Background] Xu T, Hu C, Zhu G, He X, Wu Y, Ying H. Preliminary results of a phase III randomized study comparing chemotherapy neoadjuvantly or concurrently with radiotherapy for locoregionally advanced nasopharyngeal carcinoma. Med Oncol. 2012 Mar;29(1):272-8. doi: 10.1007/s12032-010-9803-x. Epub 2011 Jan 30. PMID 21279704